CLINICAL TRIAL: NCT03923374
Title: Effects of Opioid Use Disorder in Pregnancy in Long-Term Maternal/Infant Outcomes
Brief Title: Opioid Use Disorder in Pregnancy in Long-Term Maternal/Infant Outcomes
Acronym: Mother/BabyOUD
Status: Recruiting | Type: Observational
Sponsor: Senthil Sadhasivam (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Senthil Sadhasivam, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY21110112; 1R01HD096800-01 (NIH)
Record Dates: First submitted 2018-10-24; First posted 2019-04-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Opioid-use Disorder; Opioid Use, Unspecified; Buprenorphine Dependence
Keywords: Pregnant with Opioid Use Disorder; Opioid Use Disorder ( OUD); Subutex; Buprenorphine; Pregnant taking buprenorphine/subutex
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Collection of DNA/Genetic/Epigenetic Samples from the mother at enrollment, then the infant at birth.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Mothers with Opioid Use Disorder: Planned recruitment of 200 pregnant (<16weeks) mothers who have opioid use disorder and are taking buprenorphine
  Interventions: Drug: Subutex / Buprenorphine; Diagnostic Test: Fetal & Neonatal MRI; Diagnostic Test: DNA/Genetic/Pharmacokenetic Blood Draws
- Pregnant Mothers: Planned recruitment of 100 pregnant (>16weeks) mothers who do not have any history of opioid use disorder.
  Interventions: Diagnostic Test: Fetal & Neonatal MRI; Diagnostic Test: DNA/Genetic/Pharmacokenetic Blood Draws

INTERVENTIONS:
Drug: Subutex / Buprenorphine — Pregnant Mothers must be taking buprenorphine / subutex for opioid use disorder.
  Groups: Pregnant Mothers with Opioid Use Disorder
Diagnostic Test: Fetal & Neonatal MRI — Mothers who consent will be given a fetal MRI and after the baby is born, a neonatal MRI.
Diagnostic Test: DNA/Genetic/Pharmacokenetic Blood Draws — Throughout the pregnancy, Mothers will be participating in blood collection throughout the study. At enrollment, we will collect DNA, Genetic and PK blood specimens, then throughout the study, we will be collecting random PK samples.

SUMMARY:
The objective of this study is to better understand the comprehensive integration of both clinical and genetic factors that will help to identify mothers who could be at an increased risk of poor response to opioid substitution and infants at risk of significant neonatal abstinence syndrome (NAS).

DETAILED DESCRIPTION:
One of the greatest impacts on maternal/infant health in the United States today is mother's who have opioid use disorder also known as OUD. This study will look at how in-utero buprenorphine also known as subutex, effects both mother/fetus in prenatal stages with MRI's, blood draws, and a series of assessments. After the neonate is born, there will be follow-up with that baby for up to 2 years with another neonatal MRI, blood draws and infant/child assessments. Planning to enroll 200 mothers who have opioid use disorder and 100 mothers with no previous opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Age greater 18 years
* Currently taking Buprenorphine for Opioid Use Disorder and enrolled in a prenatal opioid maintenance program in the antenatal clinic at IU Health University Hospital.
* Pregnant with single baby
* Planned delivery at Methodist, University or Riley Hospital

Exclusion Criteria:

* Serious maternal medical illness as deemed by study physician or investigator.
* Known or suspected major fetal/neonatal congenital abnormalities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any woman of the age of 18 or older that is having a single pregnancy, and currently taking buprenorphine for opioid use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of opioid misuse severity using assessments | 5 years
  Incidence of opioid misuse severity and buprenorphine treatment response will be assessed by the treating physician using assessments such as Who Assist, TCU Motform, Adverse Childhood Experience Assessment, Ham-A and Ham-D.
Pharmacological treatment for neonatal abstinence syndrome | 5 years
  Incidence of Neonatal Abstinence Syndrome and need for pharmacological treatment.

SECONDARY OUTCOMES:
Incidence of adverse effects of buprenorphine using MRI | 5 years
  Incidence of adverse effects of buprenorphine use on fetal and placental changes using MRI.
Concentration of long-term neurodevelopmental outcomes using assessments | 5 years
  Concentration of long-term neurodevelopmental outcomes in neonates using the Ages and Stages Questionnaire and the Baileys follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Senthil Sadhasivam, MD, MPH, Principal Investigator — University of Pittsburgh, UPMC
Locations (1):
- UPMC Children's Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided